CLINICAL TRIAL: NCT01016951
Title: A Phase I, Multi Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of AZD9164 Given Once Daily as Inhaled Formulation Via Turbuhaler for 13 Days in Healthy Male and Female Subjects and in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Multiple Ascending Dose Study With AZD9164 Given for 13 Days in Healthy Male and Female Subjects and in Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped since it was considered that one of the pre-defined stopping criterion was met.
Sponsor: AstraZeneca (Industry)
Responsible Party: Carin Jorup MD, Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1882C00002; EudraCT number: 2009-015645-23
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Healthy; COPD
Keywords: Phase I; Safety study; AZD9164
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD9164
  Interventions: Drug: AZD9164 Turbuhaler®
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Turbuhaler®

INTERVENTIONS:
Drug: AZD9164 Turbuhaler® — Dry powder for inhalation via Turbuhaler, MAD. Starting dose in healthy volunteers is 400 µg with up to two dose escalations not exceeding AstraZeneca pre-defined exposure limits.
  The COPD patients will receive a dose of 1000 µg.
  Arms: A
Drug: Placebo Turbuhaler® — Dry powder for inhalation via Turbuhaler, MAD
  Arms: B

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of inhaled AZD9164 following administration of multiple ascending doses in healthy male and female subjects and COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female, age 18-45, COPD patients > 40 years
* Healthy subjects and COPD patients; Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy subjects; Females must have a negative pregnancy test, must not be lactating and must be of non-child-bearing potential, by the following criteria: - irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy
* COPD patients; Females must have a negative pregnancy test, must not be lactating and must be of non-child-bearing potential, by the following criteria: Post menopausal. Woman below 50 years old will be considered post menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments, and with LH and FSH levels in the post menopausal range. Women over 50 years of age will be considered post menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment. - irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy
* Healthy subjects; Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg
* COPD patients; Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Healthy subjects; Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results of the subject's ability to participate in the study
* COPD patients; Any clinically significant disease or disorder (other than COPD) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results of the subject's ability to participate in the study
* Healthy subject and COPD patients; Any clinically significant abnormalities in clinical chemistry, haematology, urinalysis or physical examination results as judged by the investigator
* Healthy subject and COPD patients; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety measurements (ECG's, Telemetry, Pulse, Blood Pressure, Safety Laboratory and Adverse Events) | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study

SECONDARY OUTCOMES:
Pharmacokinetics samples for AZD9164 | PK sampling during the residential period and intense PK sampling day 1 and 15 in healthy and day 13 in COPD patients
Investigation of PD effects | Spirometry at screening and during the residential stay

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, Study Director — AstraZeneca R&D, Lund, Sweden; Aslak Rautio, Principal Investigator — Quintiles Hermelinen AB
Locations (2):
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Luleå

REFERENCES:
- [Derived] Jorup C, Bengtsson T, Strandgarden K, Sjobring U. Transient paradoxical bronchospasm associated with inhalation of the LAMA AZD9164: analysis of two Phase I, randomised, double-blind, placebo-controlled studies. BMC Pulm Med. 2014 Mar 27;14:52. doi: 10.1186/1471-2466-14-52. PMID 24669829